CLINICAL TRIAL: NCT05995847
Title: The Effectiveness of Harmonica Playing in Improving Lung Function Among In-home Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effectiveness of Harmonica Playing in Improving Lung Function Among COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zeng Qiuxuan, nurse-in-charge, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZQiuxuan
Record Dates: First submitted 2023-07-03; First posted 2023-08-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- harmonica combination group (Experimental): These patients will participate in a six-month harmonica playing program, in addition to receiving basic pulmonary rehabilitation (PR) care, which includes self-management education, exercise training, and breathing training, as well as routine follow-up. All training sessions are home-based and will take place five days per week for six months.
  Interventions: Behavioral: Harmonica playing program plus basic PR care with routine follow-up
- basic-PR-care group (Active Comparator): These patients will receive basic pulmonary rehabilitation (PR) care, which includes self-management education, exercise training, and breathing training, as well as routine follow-up. All training sessions are home-based and will take place five days per week for six months.
  Interventions: Behavioral: Basic PR care with routine follow-up

INTERVENTIONS:
Behavioral: Harmonica playing program plus basic PR care with routine follow-up — The intervention will last for a total of six months. During this period, patients are expected to play the harmonica daily for 30 minutes, five days a week. Additionally, patients will receive basic pulmonary rehabilitation (PR) care, which includes self-management education, exercise training, and breathing training, as well as routine follow-up. All training sessions are home-based and will take place five days per week for the duration of six months.
  Arms: harmonica combination group
Behavioral: Basic PR care with routine follow-up — These patients will receive basic pulmonary rehabilitation (PR) care, which includes self-management education, exercise training, and breathing training, as well as routine follow-up. All training sessions are home-based and will take place five days per week for the duration of six months
  Arms: basic-PR-care group

SUMMARY:
Although it has been documented that harmonica playing plays a role in the pulmonary rehabilitation (PR) of patients with chronic obstructive pulmonary disease (COPD), current studies are limited by small sample sizes, uncomprehensive outcome indicators, and short intervention durations. Thus, the investigators aim to compare the harmonica combination group with the basic-PR-care group in terms of improving health outcomes among COPD patients, such as lung function, self-efficacy, quality of life, compliance with training, and emotional distress.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is an avoidable and treatable condition characterized by chronic respiratory symptoms and airflow obstruction, primarily due to airway and/or alveolar abnormalities from toxic elements. Because of COPD's high prevalence and mortality, its prevention and treatment pose a global public health challenge that needs addressing.

Pulmonary rehabilitation (PR) is considered a cornerstone of COPD management because it effectively improves exercise tolerance, exercise-induced dyspnea, fatigue, and health-related quality of life. Inspiratory muscle training (IMT) plays an important role in PR. Studies suggest that harmonica playing can emulate inspiratory muscle training, enhancing pulmonary function in COPD patients. Additionally, as a music therapy approach, harmonica playing may alleviate the emotional distress often seen in these individuals.

However, existing studies haven't provided robust evidence to support harmonica playing's efficacy in enhancing COPD patients' health outcomes due to limitations like small sample sizes, non-trial study designs, incomplete outcomes, and short intervention durations. It remains unclear whether harmonica playing can improve COPD patients' physiological and psychological health outcomes.

This study's primary aim is to evaluate whether harmonica playing can boost the lung function of COPD patients compared to those only receiving basic PR care in the control group. The secondary aim is to investigate if harmonica playing can enhance other outcomes related to physical and psychological aspects, such as self-efficacy, quality of life, training compliance, and emotional distress.

Methods:

This is a single-center RCT with a low-risk intervention.

Patients who meet the inclusion criteria and do not meet any exclusion criteria will be randomly assigned to either the intervention or control group. The intervention group will receive a harmonica playing program in addition to basic PR care, excluding the pursed-lip breathing exercise, along with routine follow-up. In contrast, the control group will receive basic PR care, which includes the pursed-lip breathing exercise, along with routine follow-up.

Details of the treatments in both groups are provided in the intervention section.

At baseline and six months post-intervention, the investigators will collect clinical evaluations including:

Lung function (Pulmonary function laboratory tests will be performed only at baseline and six months post-intervention) Physical activity Symptoms Quality of life Psychological well-being (focusing on depression and anxiety) Self-efficacy Fatigue Self-reported compliance and satisfaction Outcome measures will be detailed in the subsequent section.

FEV1% predicted is a commonly used outcome indicator in PR and is suitable for sample size estimation. According to results from similar studies, the minimum clinically important difference (MCID) for FEV1% predicted is 4%, with a baseline standard deviation (SD) of 10%. Given a two-tailed significance level of 0.05 and a power of 80%, each group requires a minimum of 99 participants. Accounting for a drop-out rate of 20%, an estimated 248 patients (124 per group) will be enrolled.

Statistical evaluation will be performed using the SPSS 21.0 program. The intention-to-treat (ITT) approach will be adopted for data analysis.

ELIGIBILITY:
Inclusion Criteria:

● Clinical diagnosis of COPD.

Exclusion Criteria:

* Individuals with a history of COPD exacerbation within the last 6 weeks. An exacerbation is defined as a deterioration in at least two respiratory symptoms that necessitate hospitalization.
* Individuals with comorbidities that affect physical activity, such as severe cardiac or neurological disorders, cancer, or musculoskeletal problems.
* Individuals with cognitive disorders.
* Individuals unable to speak or understand spoken/written Chinese.
* Individuals who have participated in pulmonary rehabilitation (or any other structured, disease-related physical training) within the previous 6 months.
* Individuals who have played the harmonica, or other similar instrument, regularly in the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 % predicted | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The investigators will assess patients' lung function using a lung function detector to obtain the outcome of FEV1 % predicted.

SECONDARY OUTCOMES:
Change in individual strength | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The CIS-Fatigue Scale will be used to assess the level of individual fatigue. The total score for the CIS-Fatigue can range from 7 to 56. A higher score indicates a lower level of individual strength.
Change in fatigue | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The FACIT-F scale will be used to assess changes in fatigue. The total score for the FACIT-F scale can range from 0 to 52. A higher score indicates a higher level of fatigue.
Compliance and satisfaction | After 6 months of intervention
  A self-designed questionnaire will be utilized, which contains questions about participants' compliance and satisfaction.
Change in self-efficacy | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The Chinese version of the COPD Self-Efficacy Scale for Chronic (CSES) will be employed to evaluate patients' disease self-efficacy. This is a 31-item scale, with responses ranging from 1 (not confident at all) to 5 (very confident). Responses are summed to produce a total score for each participant. Scores can range from 31 to 155, with higher scores indicating greater self-efficacy.
Change in psychological well-being | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess patients' anxiety and depression. Higher scores indicate increased levels of anxiety or depression. Subscale scores of ≥11 are considered indicative of a 'definite case'. Scores of 8 to 10 suggest a 'suspicious case', and scores of 0 to 7 are deemed a 'noncase' for anxiety or depression.
Change in quality of life | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The St. George's Respiratory Questionnaire (SGRQ) will be used to assess patients' quality of life. The total score ranges from 0 to 100. A score of 0 indicates no impairment in quality of life, while a score of 100 denotes maximum impairment. A higher score indicates a poorer quality of life.
Change in symptoms | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The COPD Assessment Test (CAT) will be employed to assess participants' symptom changes. The total score can range from 0 to 40. A higher score on the CAT indicates a more severe impact of COPD on a patient's health status and thus worse outcomes.
Change in level of physical activity | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The 6-minute walk distance, which represents the level of physical activity, will be assessed using a 6-minute walk test. A shorter 6MWD typically indicates poorer exercise tolerance and correlates with more severe disease.
Changes in levels of breathlessness | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The Modified Medical Research Council (mMRC) Dyspnea Scale will be used to gauge participants' level of breathlessness. Scores range from 0 to 4, with a higher score signifying more severe breathlessness.
Changes in clinical control | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The Clinical COPD Questionnaire (CCQ) will be utilized to gauge clinical control in participants. Total scores range from 0 to 6, with a higher CCQ score signifying poorer clinical control and a worse health status.
Social support status | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The Multidimensional Scale of Perceived Social Support (MSPSS) will be used for assess social support. The scores can range from 12 and 84. A higher score indicates greater perceived social support
Change in inspiratory muscle strength | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The investigators will assess patients' inspirtaory muscle strength using a lung function detector.
Change in expiratory muscle strength | At baseline, after 1 month, after 3 months, and after 6 months of intervention
  The investigators will assess patients' expiratory muscle strength using a lung function detector.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The first affiliated hospital of Guangzhou Medical Univeristy, Guangzhou

REFERENCES:
- [Derived] Chen W, Huang J, Zeng Q, Ye ZJ, Li J, Li J. Patient perspectives on harmonica playing as an intervention for chronic obstructive pulmonary disease: a qualitative study. BMJ Open. 2026 Feb 6;16(2):e112115. doi: 10.1136/bmjopen-2025-112115. PMID 41651516
- [Derived] Zeng Q, Lin X, Chen W, Fong DYT, Li J, Li J. Effectiveness of a harmonica-integrated, tele-supervised home-based pulmonary rehabilitation program on lung function and comprehensive health outcomes in patients with chronic obstructive pulmonary disease: a randomized controlled trial protocol. Front Public Health. 2025 Jan 29;13:1541866. doi: 10.3389/fpubh.2025.1541866. eCollection 2025. PMID 39944075